CLINICAL TRIAL: NCT05785962
Title: Electromyographic Control of the Response in the Application of Vojta Therapy in People With Brain Injury.
Acronym: ElectroVojta
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not funding
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Ana María Martín Nogueras, Principal Investigator. University Professor. Dra. Ana María Martín Nogueras, University of Salamanca
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ElectroVojta
Record Dates: First submitted 2023-03-09; First posted 2023-03-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Abdominal Muscles

STUDY DESIGN:
Intervention Model Description: Subjects in each group will be matched by age and sex.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group for people with brain damage (Experimental): Other: Vojta The subject will be placed on a stretcher with the torso uncovered. Once the adhesive electrodes have been placed in the different recording areas on the anterior part of the trunk, a recording of the activity at rest will begin, two minutes of stimulation (digital pressure), one minute of rest, two minutes of stimulation in the contralateral side and, finally, one minute of rest.
  The therapy consists of the application of a stimulating pressure in the pectoral area in the pattern of the locomotion complex of reflex rolling in its first phase. For this, the subject will be placed in a supine position aligned with respect to the axial axis, with the arms along the body, the lower extremities in extension, and the head extended with a rotation of approximately 30º towards one side of the stimulation. The manual stimulation pressure will be exerted in the space between the 6th-7th or the 7th-8th rib under the mammillary line, with a force of about 2 kg.
  Interventions: Other: Vojta Therapy
- Intervention group for people without brain damage (Experimental): Other: Vojta The subject will be placed on a stretcher with the torso uncovered. Once the adhesive electrodes have been placed in the different recording areas on the anterior part of the trunk, a recording of the activity at rest will begin, two minutes of stimulation (digital pressure), one minute of rest, two minutes of stimulation in the contralateral side and, finally, one minute of rest.
  The therapy consists of the application of a stimulating pressure in the pectoral area in the pattern of the locomotion complex of reflex rolling in its first phase. For this, the subject will be placed in a supine position aligned with respect to the axial axis, with the arms along the body, the lower extremities in extension, and the head extended with a rotation of approximately 30º towards one side of the stimulation. The manual stimulation pressure will be exerted in the space between the 6th-7th or the 7th-8th rib under the mammillary line, with a force of about 2 kg.
  Interventions: Other: Vojta Therapy

INTERVENTIONS:
Other: Vojta Therapy — The therapy consists of the application of a stimulating pressure in the pectoral area in the pattern of the locomotion complex of reflex rolling in its first phase. For this, the subject will be placed in a supine position aligned with respect to the axial axis, with the arms along the body, the lower extremities in extension, and the head extended with a rotation of approximately 30º towards one side of the stimulation. The manual stimulation pressure will be exerted in the space between the 6th-7th or the 7th-8th rib under the mammillary line, with a force of about 2 kg.

SUMMARY:
A non-randomized clinical trial on a cohort of healthy subjects of legal age, both sexes, recruited from the university community and who will be randomly distributed into two groups (experimental and control). The objective will be to determine the feasibility of the standardized intervention protocol on the stabilizing muscles of the trunk (external oblique and internal oblique) before, during and after the application of Vojta Therapy, and to know the effects produced on the Musculature studied after performing the intervention.

ELIGIBILITY:
Brain injury group

Inclusion Criteria :

* Over 18 and under 80 years of age
* Persons with a medical diagnosis of brain damage secondary to stroke
* Have preserved the ability to walk, even with some type of orthopedic some type of orthopedic aid,

Exclusion Criteria:

* Over 80 years
* Healthy people

Group without brain damage

Inclusion Criteria :

* Over 18 and under 80 years of age
* Healthy people
* Full cognitive capacity.

Exclusion Criteria:

* Subjects with neuro-muscular pathologies that affect the abdominal muscles, previous surgeries in the area or any chronic neurological or organic disorder that may alter the results.
* Fever

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity in abdominal muscles | Change from Baseline electromyographic activity at 10 minutes.
  The electromyographic activity of internal and external obliques in nanovolts will be collected before, during and after the intervention. Acquired signals are sampled at 1 KHz and filtered with a 60 Hz high pass digital filter to reject signals of non-muscular origin. The degree of muscle activation measured in micro volts (uV) will be recorded.

SECONDARY OUTCOMES:
Date of birth | Baseline
  It will be registered at the beginning of the study in order to calculate the age of the participant.
Sex | Baseline
  It will be registered at the beginning of the study.
Height | Baseline
  It will be registered at the beginning of the study in centimeters.
Weight | Baseline
  It will be registered at the beginning of the study in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- USAL, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No